CLINICAL TRIAL: NCT02211508
Title: A Double-Blinded, Randomized, Sham-Controlled, Pivotal Study of the NeuroPoint Device for the Treatment of Pain Associated With Fibromyalgia
Brief Title: Prospective Evaluation of RINCE to Reduce Fibromyalgia Effects - 301
Acronym: PERRFECT-301
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial terminated Feb '15. Interim analysis results missed primary endpoint, intended signal not delivered in Tx arm, sham results as expected. No safety issues.
Sponsor: Cerephex Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NPT-301
Record Dates: First submitted 2014-08-06; First posted 2014-08-07 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; pain; stimulation
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12-week RINCE (Active Comparator): RINCE - active RINCE therapy involving 24 total treatment applications from NeuroPoint device
  Interventions: Device: RINCE
- Sham RINCE (Sham Comparator): Sham RINCE - sham RINCE therapy involving 24 total sham applications from NeuroPoint device
  Interventions: Device: RINCE

INTERVENTIONS:
Device: RINCE — The NeuroPoint device is used to deliver repeat applications of RINCE therapy
  Other Names: RINCE therapy; RINCE therapy delivered by the NeuroPoint device

SUMMARY:
The purpose of this study is to test the safety and efficacy of a noninvasive cortical electrostimulation therapy known as "Reduced Impedance Noninvasive Cortical Electrostimulation" (RINCE) in the treatment of pain associated with fibromyalgia. Patients who meet the 2010 American College of Rheumatology criteria for fibromyalgia will receive up to 24 RINCE treatments delivered by a medical device called "NeuroPoint". Approximately 200 fibromyalgia patients will be randomized into one of two study groups. One of these groups will receive sham treatment, meaning they will receive no treatment at all, while the other group will receive active RINCE treatment. The study's primary outcome measure will be the difference between active and sham treatment groups in the mean change from baseline in patients' weekly worst pain scores. The study's hypothesis is that there will be a difference between treatment groups in primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female, 22 to 65 years of age, inclusive.
* Patient has a diagnosis of primary fibromyalgia as defined by the 2010 American College of Rheumatology Preliminary Diagnostic Criteria for fibromyalgia.
* If female, is either not of childbearing potential or is willing to utilize specified practices throughout the study to prevent becoming pregnant.
* Patient is willing and able to refrain or withdraw from the following therapies for the duration of the study: duloxetine, milnacipran, pregabalin, gabapentin, naltrexone, sodium oxybate, and opiates.
* Qualified patients with mild or moderate depression must be clinically stable, without risk of suicidal ideation or behavior, and the dose of allowed anti-depressants should have been stable for at least three months prior to the Baseline clinic visit.
* Patient is willing and able to comply with all protocol-specified requirements.
* Patient is capable of reading and understanding English and has provided written informed consent to participate.

Exclusion Criteria:

* The patient suffers from one or more of clinically significant psychiatric condition that could interfere with the patient's well-being or ability to comply with the protocol.
* Patient has a Beck Depression Inventory-II total score greater than 25 at either the Screening visit or Baseline clinic visit.
* The patient is at increased risk of suicide.
* Patient is unable, unwilling or not advised to refrain from or discontinue prohibited medications or treatments.
* Patient has a diagnosis of, or is being treated for, systemic lupus erythematosus, inflammatory arthritis, or other documented systemic autoimmune disorder, Parkinson's disease, multiple sclerosis, or cancer (other than basal or squamous cell skin cancer).
* Patient has any other chronic pain condition that, in the Investigator's or Sponsor's opinion, could interfere with the patient's assessment of his/her fibromyalgia status.
* Patient has a history of severe, refractory or uncontrolled migraine headaches, seizure disorder or clinically significant cognitive dysfunction.
* Patient is pregnant or planning to become pregnant within the next 6 months.
* Patient has a body mass index greater than 40 at the Screening visit.
* Patient has a history of cranial electrical stimulation or transcutaneous magnetic stimulation within 2 years of screening, or electroconvulsive therapy within 5 years of screening.
* Patient has a metal implant at or above the level of the 7th cervical vertebra, a cardiac pacemaker or defibrillator, or vagus nerve stimulator.
* Any recent surgery or anticipated need for surgery that might confound results or interfere with patient's ability to comply with the protocol.
* Myocardial infarction during the 12 months prior to screening, uncontrolled hypertension, active cardiac disease, clinically significant cardiac rhythm or conduction abnormality, or anticipation of bypass or other cardiac surgery within the next 12 months.
* Current systemic infection (e.g., HIV, hepatitis B or C; Lyme disease).
* Patient is using opiates on a regular or frequent basis.
* Pending or current litigation or disability claim (including Workman's Compensation).
* History of significant alcohol and/or drug abuse or dependency within preceding 5 years, or a positive result on the screening (or subsequent) drug screen indicating use of an illicit substance.
* Patient has participated in an investigational study of a therapeutic treatment within 90 days prior to Screening visit or is currently participating in another clinical trial.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in patients' 24-hour recall worst pain intensity | Assessed at 12 weeks
  The primary efficacy endpoint will be the contrast at 12 weeks versus Baseline in the (paired) mean weekly change in patients' self-reported daily (24-hour) recall worst pain intensity using an 11-point (0-10) numerical rating scale.

SECONDARY OUTCOMES:
Patient self-reported Global Impression of Change | Assessed at 12 weeks
Proportion of patients in the treatment and sham groups whose average daily worst pain intensity decreased by at least 50% | Assessed at 12 weeks
  Worst pain intensity evaluated using an 11-point (0-10) numerical rating scale.
Change from baseline in Revised Fibromyalgia Impact Questionnaire | Assessed at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: R. Michael Gendreau, MD PhD, Study Director — Cerephex Corporation
Locations (16):
- United States (16):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Premier Research, Phoenix, Arizona
  - Neurovations, Napa, California
  - Superior Research LLC, Sacramento, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Avail Clinical Research, DeLand, Florida
  - Compass Research LLC, Orlando, Florida
  - Chicago Research Center, Chicago, Illinois
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Fieve Clinical Research, New York, New York
  - Upstate Clinical Research Associates, Williamsville, New York
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Sunstone Medical Research, Medford, Oregon
  - Omega Medical Research, Warwick, Rhode Island
  - Fatigue Consultation Clinic, Salt Lake City, Utah
  - Swedish Clinical Research, Seattle, Washington

REFERENCES:
- [Background] Hargrove JB, Bennett RM, Simons DG, Smith SJ, Nagpal S, Deering DE. A randomized placebo-controlled study of noninvasive cortical electrostimulation in the treatment of fibromyalgia patients. Pain Med. 2012 Jan;13(1):115-24. doi: 10.1111/j.1526-4637.2011.01292.x. PMID 22233397
- [Background] Hargrove JB, Bennett RM, Clauw DJ. Long-term outcomes in fibromyalgia patients treated with noninvasive cortical electrostimulation. Arch Phys Med Rehabil. 2012 Oct;93(10):1868-71. doi: 10.1016/j.apmr.2012.04.006. Epub 2012 Apr 21. PMID 22525670